CLINICAL TRIAL: NCT00896740
Title: Analysis of Fanconi Anemia Gene Function by Microarray Analysis of Bone Marrow Cells
Brief Title: Gene Function in Bone Marrow Cells From Patients With Fanconi Anemia and From Healthy Participants
Status: Terminated | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Grover Bagby, Professor Emeritus, OHSU Knight Cancer Institute
Other Study IDs: IRB00000713; OHSU-HEM-01079-L; CDR0000445212 (Other: NCI PDQ)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Microarray Analysis; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: microarray analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with Fanconi anemia and from healthy participants in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to Fanconi anemia.

PURPOSE: This laboratory study is evaluating gene function in bone marrow cells from patients with Fanconi anemia and from healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the complete hematopoietic transcriptomes of Fanconi cells of every common complementation group (e.g., A, C, G, and F) as well as transcriptomes of neoplastic cells derived from bone marrow of patients with Fanconi anemia.
* Define large-scale dynamic gene expression data in these patients.

OUTLINE: This is a multicenter study.

Patients and healthy volunteers undergo bone marrow aspiration or biopsy for biological studies. Samples are analyzed for gene expression profiles using microarray assays.

PROJECTED ACCRUAL: A total of 80 patients and 10 healthy volunteers will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of Fanconi anemia

    * Requires bone marrow aspiration or biopsy for clinical purposes
  * Healthy volunteer

    * Over 18 years of age
    * No known blood abnormality

PATIENT CHARACTERISTICS:

* Platelet count > 150,000/mm^3
* White Blood Cell(WBC) > 4,000/mm^3
* Hemoglobin > 13 g/dL
* No clinical signs or symptoms of acute or subacute infection (e.g., viral, bacterial, or fungal)
* No allergies to lidocaine or xylocaine

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: FA Patients are recruited from OHSU Clinics. Healthy Normal donors are recruited with an IRB approved advertisement which runs in the Outlook and is posted on bulletin boards around campus
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2002-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Fanconi anemia (FA) hematopoietic cells vs normal hematopoietic cells
Comparison of FA hematopoietic cells from children with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) vs children (siblings) with FA but without MDS/AML
Comparison of FA cells from different complementation groups

CONTACTS AND LOCATIONS:
Overall Officials: Grover C. Bagby, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States